CLINICAL TRIAL: NCT02654613
Title: Addressing Challenges in Scaling up TB and HIV Treatment Integration in Public Health Settings in South Africa
Brief Title: Scaling up TB and HIV Treatment Integration
Acronym: SUTHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: BroadReach Healthcare (Industry); Institute for Healthcare Improvement (Other)
Responsible Party: Principal Investigator, Dr Kogieleum Naidoo, Dr, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CAP013
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: HIV; Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quality Improvement Intervention (Active Comparator): In intervention clinics, staff will follow QI methodology to undertake a detailed assessment of their HIV-TB care and to prioritize the steps to improve treatment outcomes. A senior nurse will be identified to be the QI champion and will be trained by the study team to fulfil this role. The QI champion in the clinic then provides peer-leadership, mentorship and support for the implementation of the prioritized changes until the checklist is complete and all integrated HIV-TB service components meet the required standard.
  Interventions: Other: Quality Improvement Model of Care
- Control Standard of Care (No Intervention): The control arm will continue with the usual support that is received for HIV-TB service integration

INTERVENTIONS:
Other: Quality Improvement Model of Care — QI addresses the "how" of program implementation. Technically, QI improves process performance by developing a common simplified view of the components and linkages of integrated care, real-time data feed-back to track system performance, understanding the psychology of system change, and crucially, the iterative testing and incorporation of ideas for performance improvement from the front-line practitioners, managers, and customers in the local context.
  Arms: Quality Improvement Intervention

SUMMARY:
This study addresses the highest ranking health research priority in South Africa, which is, to develop and test optimal models of HIV-TB service delivery that will enhance retention, adherence and coverage of HIV-TB co-infected patients. HIV and TB are highest in sub-Saharan Africa, a region with limited health budgets, infrastructure, human resources, and suboptimal TB infection control practices. There is compelling clinical evidence suggesting that integrating HIV and TB services saves lives and presents an effective and efficient use of resources directed at optimizing health outcomes. Quality improvement (QI) methods are increasingly being used to systematically test and incorporate local ideas into strategies for reliable implementation and scale up. This trial is designed to test a practical, implementable and affordable strategy aimed at improving HIV-TB service integration to reduce TB and HIV associated deaths. This is a cluster randomized controlled trial, which evaluates and tests the effectiveness of implementing a QI model to integrate HIV-TB service delivery in primary health care clinics, on reducing morbidity and mortality in TB-HIV co-infected patients. This study will be conducted in 2 districts, Ugu and uThungulu, in KwaZulu-Natal, South Africa. The model of integrated care delivery for TB and HIV using the QI method offers a systems approach to care delivery to directly enhance treatment outcomes by enabling comprehensive effective care designed around the patients journey from entry to the clinic, through screening treatment initiation, treatment completion, and retention in care that is directed at the goals of cure for TB, effective sustainable HIV viral suppression and reduced HIV associated TB mortality as the main health impact. The scalability of the model, once proven effective, is the critical element that makes it increase population coverage of quality diagnosis and treatment of HIV-TB co-infection. QI methods promote front line staff engagement in identification and rapid testing of local implementation solutions to gaps in performance of processes of care along the steps of the patient journey. Gaps in care are identified through continuous feedback on a core set of indicators collected monthly as routine collection of data.

DETAILED DESCRIPTION:
The primary aim of this study is to test the effectiveness of a peer mentor-led, quality-improvement model of service delivery of integrated HIV-TB treatment on mortality in HIV-TB co-infected patients treated in rural primary health care clinics in KwaZulu-Natal, South Africa

Specific Objectives (i) To determine the impact of a QI-mediated HIV-TB service integration on patient mortality. All patients that access services in intervention and control clinics, via either the TB entry point or via the HIV entry point will be tracked during clinic follow-up visits or, through a community care giver, and will have their vital status ascertained 12 months after clinic randomization.

(ii) To determine the effectiveness of peer-led Quality Improvement (QI) to integrate HIV-TB services. The effect, on HIV-TB integrated processes of care, of the deployment of a QI approach (systems view, data driven decision making, culture of continuous improvement, trained peer mentors) to ensure uniform implementation of an essential package of evidence based HIV-TB interventions that support HIV-TB integration. The impact on clinical outcomes of using QI methods to implement integrated HIV and TB management will be assessed using the following indicators: Time to ART initiation among HIV infected TB suspects and cases; HIV testing rates in TB patients; Number of HIV-TB co-infected patients receiving co-treatment for TB and HIV at the same facility; Number of patients infected with HIV or TB that are retained in care at 12 months; Indicators of treatment adherence such as - number of HIV patients that are virologically suppressed at 12 months and TB treatment outcomes; Hospitalisation rates among patients receiving co-treatment for TB and HIV.

(iii) To identify clinic-level factors that impact on integrated HIV-TB services. Understanding the context (environmental, social and political factors) in which we are working is essential to identifying factors that promote or inhibit the implementation of the intervention. We will use the COACH tool (Context Assessment for Community Health) [8] to collect data and assess the organizational context and the influence of factors such as organizational culture, leadership, resources and HCWs remuneration etc. on the intervention

(iv) To determine the cost-effectiveness of implementing HIV-TB services using Quality Improvement methodology (Intervention Clinics) versus the base-case of implementing HIV-TB services independently, through a within-trial approach using both health service (e.g. training, remuneration) and patient costs (e.g. travel, opportunity costs) as inputs. We will also calculate total intervention costs to assess its affordability and explore cost-effectiveness under various scenarios (e.g. different TB-HIV co-infection rates) using decision analytical modeling.

(v) To identify a set of interventions, change ideas, tools and approaches that can be used to scale up adoption, implementation and sustainability of integrated HIV-TB services across South Africa and in other resource constrained settings.

(vi) To strengthen the capacity of CAPRISA to independently perform implementation research in PRDs, including community-randomized trials and health economic analysis, through expert mentoring and supervision of PhD programmes.

ELIGIBILITY:
Inclusion Criteria:

* South African Department of Health Primary Health Care Clinics
* ART site
* Supported by BroadReach Healthcare

Exclusion Criteria:

* Mobile clinics
* Clinics that do not offer ART
* Clinics with only 1 nurse
* Hospitals and Gateway clinics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 12 months
  Mortality rate in TB-HIV co-infected patients

SECONDARY OUTCOMES:
HIV testing rates | 12 months
  HIV testing rates in TB patients
Intensified Case Finding for TB | 12 Months
  TB Screening in HIV infected patients
Cotrimoxazole for HIV-TB patients | 12 months
  Initiating Cotrimoxazole in HIV-TB patients
Retention in HIV-TB patients | 12 months
  Enhanced retention in care strategies including the use of community care workers for retention and for community based management of selected patients
ART initiation in HIV-TB co-infected patients | 12 months
  Initiating ART in co-infected patients irrespective of CD4 count
Integrated Data Management System | 12 months
  1 data management system for co-infected patients , including 1 file , 1 appointment and 1 health care worker addressing both HIV and TB care and treatment
HIV and TB Adherence Strategy | 12 months
  • Enhanced ART and TB treatment adherence strategies including the use of community care workers for adherence support and for community based management of selected patients

CONTACTS AND LOCATIONS:
Overall Officials: Kogieleum Naidoo, MBChB, Principal Investigator — Centre for the AIDS Programme of Research in South Africa
Locations (1):
- CAPRISA eThekwini Clinical Research Site, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naidoo K, Zuma NY, Moodley M, Made F, Perumal R, Gengiah S, Ngozo J, Padayatchi N, Nunn A, Karim SA. High mortality among patients with tuberculosis accessing primary care facilities: secondary analysis from an open-label cluster-randomised trial. EClinicalMedicine. 2025 Mar 18;82:103151. doi: 10.1016/j.eclinm.2025.103151. eCollection 2025 Apr. PMID 40166654
- [Derived] Naidoo K, Gengiah S, Yende-Zuma N, Mlobeli R, Ngozo J, Memela N, Padayatchi N, Barker P, Nunn A, Karim SSA. Mortality in HIV and tuberculosis patients following implementation of integrated HIV-TB treatment: Results from an open-label cluster-randomized trial. EClinicalMedicine. 2022 Feb 12;44:101298. doi: 10.1016/j.eclinm.2022.101298. eCollection 2022 Feb. PMID 35198922
- [Derived] Gengiah S, Connolly C, Yende-Zuma N, Barker PM, Nunn AJ, Padayatchi N, Taylor M, Loveday M, Naidoo K. Organizational contextual factors that predict success of a quality improvement collaborative approach to enhance integrated HIV-tuberculosis services: a sub-study of the Scaling up TB/HIV Integration trial. Implement Sci. 2021 Sep 17;16(1):88. doi: 10.1186/s13012-021-01155-7. PMID 34535170
- [Derived] Gengiah S, Barker PM, Yende-Zuma N, Mbatha M, Naidoo S, Taylor M, Loveday M, Mhlongo M, Jackson C, Nunn AJ, Padayatchi N, Karim SSA, Naidoo K. A cluster-randomized controlled trial to improve the quality of integrated HIV-tuberculosis services in primary healthcareclinics in South Africa. J Int AIDS Soc. 2021 Sep;24(9):e25803. doi: 10.1002/jia2.25803. PMID 34498370
- [Derived] Naidoo K, Gengiah S, Yende-Zuma N, Padayatchi N, Barker P, Nunn A, Subrayen P, Abdool Karim SS. Addressing challenges in scaling up TB and HIV treatment integration in rural primary healthcare clinics in South Africa (SUTHI): a cluster randomized controlled trial protocol. Implement Sci. 2017 Nov 13;12(1):129. doi: 10.1186/s13012-017-0661-1. PMID 29132380